CLINICAL TRIAL: NCT06009510
Title: Participation Trends in Bladder Cancer Clinical Trials - Exploring Engagement Dynamics Among Individuals Impacted by Bladder Cancer
Brief Title: Exploring Engagement Dynamics Among Individuals Impacted by Bladder Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 87986229
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Bladder Cancer
Keywords: bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study seeks to delve into the firsthand experiences of patients diagnosed with bladder cancer who partake in a separate clinical trial featuring a specific medical intervention. The primary emphasis will be on meticulously tracking the rates of trial completion and withdrawal among these individuals.

By joining this clinical trial, individuals have the unique opportunity to contribute to the betterment of future bladder cancer patients and play an active role in advancing medical research.

ELIGIBILITY:
Inclusion Criteria:

* Patient has self-identified as planning to enroll in a clinical trial
* Patient has been diagnosed with bladder cancer
* Patient is a minimum of 18 years or older

Exclusion Criteria:

* Patient does not understand, sign, and return consent form
* Inability to perform regular electronic reporting
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bladder cancer patients who are actively considering enrolling in an observational clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to participate in a bladder cancer clinical research | 3 months
Rate of patients who remain in bladder cancer clinical research to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ng K, Stenzl A, Sharma A, Vasdev N. Urinary biomarkers in bladder cancer: A review of the current landscape and future directions. Urol Oncol. 2021 Jan;39(1):41-51. doi: 10.1016/j.urolonc.2020.08.016. Epub 2020 Sep 9. PMID 32919875
- [Background] Gaya JM, Territo A, Woldu S, Schwartzmann I, Verri P, Gonzalez-Perez L, Cozar JM, Minana B, Medina RA, de la Rosa-Kehrmann F, Lozano-Palacio F, Ribal MJ, Hernandez C, Castineiras JJ, Requena MJ, Moreno J, Caraballido JA, Baena V, Breda A, Palou Redorta J. Incidental diagnosis of bladder cancer in a national observational study in spain. Actas Urol Esp (Engl Ed). 2023 Jun;47(5):296-302. doi: 10.1016/j.acuroe.2022.09.005. Epub 2022 Oct 1. English, Spanish. PMID 36443223
- [Background] Malhotra B, Hiteshi P, Khalkho P, Malik R, Bhadada SK, Bhansali A, Shafiq N, Malhotra S, Kumar N, Rajput R, Rastogi A. Bladder cancer with pioglitazone: A case-control study. Diabetes Metab Syndr. 2022 Nov;16(11):102637. doi: 10.1016/j.dsx.2022.102637. Epub 2022 Oct 8. PMID 36270237

DOCUMENTS (1):
  • Informed Consent Form (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT06009510/ICF_000.pdf